CLINICAL TRIAL: NCT05788835
Title: Drug-eluting Bead Transarterial Chemoembolization and Drug-eluting Bead Transarterial Chemoembolization Sequential Hepatic Artery Chemotherapy Infusion for Unresectable BCLC Stage C HCC: A Randomized Controlled Trial
Brief Title: DEB-TACE Versus DEB-TACE Sequential HAIC for Unresectable BCLC Stage C HCC; A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuhua Duan (Other)
Responsible Party: Sponsor-Investigator, Xuhua Duan, Associate Professor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY-0081-002
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: HCC
Keywords: DEB-TACE- HAIC; DEB-TACE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB-TACE-HAIC (Experimental): Drug-eluting bead transarterial chemoembolization Sequential with FOLFOX-based chemotherapy hepatic artery infusion
  Interventions: Procedure: DEB-TACE and HAIC
- DEB-TACE (Active Comparator): Drug-eluting bead transarterial chemoembolization
  Interventions: Procedure: DEB-TACE

INTERVENTIONS:
Procedure: DEB-TACE and HAIC — Drug-eluting bead transarterial chemoembolization sequential Hepatic Artery Chemotherapy Infusion
  Arms: DEB-TACE-HAIC
Procedure: DEB-TACE — Drug-eluting bead transarterial chemoembolization
  Arms: DEB-TACE

SUMMARY:
This is a randomized controlled trial to determine the efficacy and safety of DEB-TACE versus DEB-TACE sequential HAIC for unresectable BCLC stage C HCC

DETAILED DESCRIPTION:
Primary liver cancer is one of the most common malignant tumors in the world. According to the survey results of the BRIDGE study, about 64% of Chinese patients with liver cancer had BCLC stage B and stage C at the first diagnosis, and the vast majority of patients in the middle and advanced stages were no longer suitable for the first choice of surgical resection and should receive comprehensive treatment mainly consisting of local treatment and systemic treatment.

TACE is one of the most used treatments for liver cancer. At present, cTACE and DEB-TACE are mainly used. Drug-eluting beads, as new drug-carrying embolisms, have the advantages of loading chemotherapeutic drugs depending on charge and releasing drugs slowly within a certain time to improve local drug concentration. Based on the application of clinical practice, its efficacy has been well confirmed. DEB-TACE results in better tumor response and a similar safety profile than cTACE. However, for HCC at stage C of BCLC, due to the large tumor load and common portal invasion, it is difficult for a single TACE to achieve complete or partial remission, and a complete embolization is likely to increase the risk of serious complications.

Hepatic Arterial Infusion Chemotherapy is used to treat hepatic arterial infusion chemotherapy (HCC). HAIC requires chemotherapy drugs to be injected directly into the liver tumor via a percutaneous arterial cannula. HAIC drugs alone stay in the tumor for a short time, will be washed out quickly, and cannot be completely covered for tumors with external hepatic collateral circulation. However, unlike HAIC, DEB-TACE can embolize tumors to nourish arteries, rapidly lead to massive ischemic necrosis of tumors, and significantly prolong the contact time between cancer cells and chemotherapy drugs. In conclusion, the combination of DEB-TACE and HAIC can make up for the respective deficiencies of DEB-TACE and HAIC. And produce enhanced local anti-tumor effect and less AEs, especially in HCC with high tumor load.

The combination of DEB-TACE and HAIC has been well tolerated in the treatment of large liver cancer. However, most patients with BCLC stage C HCC have vascular invasion or extrahepatic metastasis, which cannot be treated surgically. Moreover, the progressive involvement of vascular invasion will eventually reduce blood flow and further deteriorate liver function, resulting in impaired liver function and poor prognosis. Therefore, we predict that the DEB-TACE sequential HAIC approach will reduce AEs while achieving good efficacy.

Therefore, based on previous studies, this study intended to select patients with unresectable primary liver cancer at stage C of BCLC in a multi-center setting, and prospectively observe the efficacy of DEB-TACE followed by FOLFOX-based HAIC in the treatment of unresectable BCLC stage C patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with unresectable HCC who strictly meet the clinical diagnostic criteria of the Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2022 Edition) or who have been confirmed by histopathology or cytology, There was at least one measurable lesion (according to the requirements of mRECIST 1.1, the spiral CT scan diameter of the measurable lesion was ≥10mm or the short diameter of enlarged lymph node was ≥15mm).
2. The sum of the diameter of single or 2-3 tumors ≥5cm. Tumor stage: Stage C of BCLC.
3. Patient age between 18 and 75，male or female.
4. ECOG 0-1.
5. Expected life span ≥ 3 months.
6. No history of severe comorbidities, such as hypertension, coronary heart disease, and mental illness, and no history of severe allergies.
7. Child-Pugh A-B.
8. HBV DNA<2000 IU/ml.
9. Women of childbearing age must undergo a pregnancy test within 7 days prior to enrollment.
10. Patients sign informed consent, good compliance, cooperate with treatment.

Exclusion Criteria:

1. Imaging examinations were conducted for HCC patients with large liver tumors (≥60% of liver volume), or carcinoma thrombus in main portal vein (occupying ≥50% of vascular diameter), or carcinoma thrombus invading mesenteric vein or inferior vena cava, or significant arteriovenous/venous fistula.
2. Before participating in this study, she had received local treatment such as TACE, external radiotherapy and radioactive particle implantation, and had undergone systemic chemotherapy, oral liver cancer targeting drugs (Sorafenib, Lenfacitinib, Apatinib) and immunotherapy such as PD-1/PD-L1/CDLA-4.
3. Diffuse liver cancer patients.
4. Patients with grade Ⅱ or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450ms for men and 470ms for women.
5. A history of gastrointestinal bleeding within the past 6 months or a definite tendency to gastrointestinal bleeding.
6. Abnormal clotting function, bleeding tendency or receiving thrombolytic or anticoagulant therapy.
7. Patients with central nervous system metastases or known brain metastases. Co-infected patients with HIV; Pregnant or lactating patients. Patients preparing for liver transplantation (other than those with previous liver transplantation.
8. Systemic failure, estimated survival time <3 months.
9. Severe renal dysfunction.
10. The patients could not complete the treatment plan due to various reasons, and lost control within three months after enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from the first DEB-TACE treatment to either radiological progression or death or up to 36 months
  Time from the first DEB-TACE treatment to either radiological progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | Time from the first DEB-TACE treatment to death or up to 36 months
  Time from the first DEB-TACE treatment to death from any cause or the end of the study
Objective response rate (ORR) | 1, 3, 6,12 months after the first DEB-TACE treatment, up to death or 36 months, whichever came first
  Proportion of patients with reduction in stable in tumor burden of a predefined amount
Disease control rate (DCR) | 1, 3, 6,12 months after the first DEB-TACE treatment, up to death or 36 months, whichever came first
  Proportion of patients with reduction or keeping in stable in tumor burden of a predefined amount
Time to Progression (TTP) | Time from the first DEB-BACE treatment to either radiological progression up to 36 months
  Time to progression was defined as the period of time from the first on-study DEB-TACE to radiographic disease progression at any site by mRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Xuhua, Ph.D., Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (16):
- China (16):
  - Luo He Central Hospital, Luohe, Henan
  - Luo Yang Central Hospital, Luoyang, Henan
  - Deng zhou People's Hospital, Nanyang, Henan
  - Nan Yang Central Hospital, Nanyang, Henan
  - General Hospital of Pingmei Shenma Group, Pingdingshan, Henan
  - First People's Hospital of Shangqiu, Shangqiu, Henan
  - Shangqiu Municipal Hospital, Shangqiu, Henan
  - Xin Yang Central Hospital, Xinyang, Henan
  - The Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Zhou Kou Central Hospital, Zhoukou, Henan
  - First People's Hospital of Zhu Madian, Zhumadian, Henan
  - Zhu Ma Dian Central Hospital, Zhumadian, Henan
  - Zhu Madian Traditional Chinese Medicine Hospital, Zhumadian, Henan
  - Second People's Hospital of Jiaozuo, Jiaozuo